CLINICAL TRIAL: NCT02325453
Title: A Multi-Institutional Chart Review to Compare the Outcomes of Robotic, Laparoscopic and Open Surgery for Gastric Cancer.
Brief Title: Robotic, Laparoscopic and Open Surgery for Gastric Cancer Compared on Surgical, Clinical and Oncological Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Study Group on Minimally Invasive Surgery for Gastric Cancer (Other)
Collaborators: Fondazione CARIT (Unknown); LOGIX S.r.l. (Unknown)
Responsible Party: Principal Investigator, Amilcare Parisi, Dr., Azienda Ospedaliera Santa Maria, Terni, Italy
Other Study IDs: 001
Record Dates: First submitted 2014-12-16; First posted 2014-12-25 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Gastric Cancer
Keywords: Robotic Surgery; Laparoscopic Surgery; Minimally Invasive Surgery; Robotic Gastrectomy; Laparoscopic Gastrectomy; Open Gastrectomy; Gastric Surgery
MeSH Terms: conditions — Stomach Neoplasms | interventions — Robotic Surgical Procedures; Laparoscopy; Conversion to Open Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Robotic Surgery: Patients underwent gastric surgery through the use of a robotic system.
  Interventions: Procedure: Robotic Surgery
- Laparoscopic Surgery: Patients underwent gastric surgery with laparoscopic procedures.
  Interventions: Procedure: Laparoscopic Surgery
- Open Surgery: Patients underwent gastric surgery with open approach.
  Interventions: Procedure: Open Surgery

INTERVENTIONS:
Procedure: Robotic Surgery — Surgical procedure performed with a robotic system.
  Groups: Robotic Surgery
Procedure: Laparoscopic Surgery — Surgical procedure performed with laparoscopic techniques.
  Groups: Laparoscopic Surgery
Procedure: Open Surgery — Traditional approach for gastric cancer.
  Groups: Open Surgery

SUMMARY:
Gastric cancer represents a great challenge for health care providers and requires a multidisciplinary context in which surgery plays a main role.

Minimally invasive surgery has been progressively developed, first with the advent of laparoscopy and more recently with the spread of robotic systems, but a number of issues are currently being debated, including the limitations in performing effective extended lymph node dissections and, in this context, the real advantages of using the robotic systems, the possible role for the Advanced Gastric Cancer, the reproducibility of completely intracorporeal techniques and the oncological results achievable during follow-up.

A multicenter study with a large number of patients is now needed to further investigate the safety and efficacy as well as long-term outcomes of robotic surgery, traditional laparoscopy and the open approach.

DETAILED DESCRIPTION:
Overall purpose:

The Overall purpose is to develop a multi-institutional database comprising information regarding surgical, clinical and oncological features of patients undergoing surgery for gastric cancer with robotic, laparoscopic or open approaches and subsequent follow-up at participating centers.

General study design:

The registry will be established by retrospectively identifying subjects with gastric cancer treated at the participating centers.

Information gathered will be obtained from existing data and records, diagnostic tests and surgical interventions.

Information will be collected and recorded by all institutes through a specific online shared system.

Main objectives:

* To determine the surgical, clinical, and oncological outcomes in both the short and long term
* To compare results according to the type of intervention, device used and manner of execution of different surgical phases
* To relate results of different surgeries with baseline characteristics of patients and stage of disease

Clinical relevance:

Studies that reported results of minimally invasive surgery for gastric cancer and recent meta-analysis emphasize the need for large trials.

A further consideration in this field regards the need of numerous patients to reach a statistical significance on surgical, clinical and oncological outcomes, in order to fully assess the effectiveness and the differences between the different surgical approaches.

At present, a multicenter registry may represent the best research tool to assess the role of minimally invasive approaches by comparing the methods with traditional open surgery.

Therefore, for this project, a large registry will be created by collecting data from the different participating centers to create a working basis for analyzing outcomes of interest and obtaining directions for further investigation.

The data collected will clarify the role of laparoscopic and robotic surgery versus the open approach in terms of:

* safety and feasibility based on the intraoperative outcomes
* respect of oncological principles in relation to the stage and location of the tumor
* recovery of gastrointestinal function considering the outcomes measured during the postoperative hospital stay
* incidence, types and severity of postoperative complications
* overall survival and disease-free survival

Duration of study:

The beginning of the trial is scheduled for January 2015. It is expected to end the chart review within one year.

Type of data collection:

In the present study, the following information will be collected:

* Patient Demographics
* Surgical Procedure details
* Tumor characteristics
* Operative findings
* Post-operative clinical findings
* Post-operative complications
* Follow-up details

Statistical analysis:

The dichotomous variables will be expressed as numbers and percentages, while continuous variables will be expressed as mean and standard deviation (SD) or median and interquartile range (minimum and maximum values).

Continuous variables, will be compared using one-way ANOVA with post hoc multiple comparison by Tukey's procedure. Pearson's χ2 test or Fisher's exact test, as appropriate, will be used for analysis of categorical data.

For each of these tests a value of alpha (α) < 0.05 will be considered statistically significant.

Potential risks and safety management:

Participation in the research registry involves the potential risks of a breach of confidentiality of the medical record information and associated privacy of the participants.

Such risks will be minimized by the use and the establishment of appropriate information technology services.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven gastric cancer
* Preoperative staging work-up performed by upper endoscopy / endoscopic ultrasound, and CT scan
* Early Gastric Cancer
* Advanced Gastric Cancer
* Patients treated with curative intent in accordance to international guidelines

Exclusion Criteria:

* Locally advanced tumor infiltrating neighboring organs
* Distant metastases: peritoneal carcinomatosis, liver metastases, distant lymph node metastases, Krukenberg tumors, involvement of other organs
* Patients with high operative risk as defined by the American Society of Anesthesiologists (ASA) score ≥4.
* History of gastric surgery
* Remnant gastric cancer
* Synchronous other major abdominal surgery
* Synchronous malignancy in other organs
* Palliative surgery cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects undergoing surgery for gastric cancer with robotic, laparoscopic or open approaches and subsequent follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Compare robotic and laparoscopic surgery with the open approach in terms of safety and feasibility. (Intraoperative complications.) | Intraoperative.
  Intraoperative complications.
Verify the respect of oncological principles through minimally invasive approaches in relation to the stage and location of the tumor by comparing results with open surgery. (Number of lymph nodes retrieved.) | Intraoperative.
  Number of lymph nodes retrieved.
Compare the three treatment arms in terms of recovery of gastrointestinal functions and physical status allowing the discharge of the patient. (Days of hospitalization after surgery until discharge.) | Assessment during an average period of 10 days after surgery.
  Days of hospitalization after surgery until discharge.
Compare the incidence, types and severity of early postoperative complications after gastrectomy by the three approaches. (Score based on the Clavien-Dindo classification system.) | Assessment during an average period of 10 days after surgery.
  Score based on the Clavien-Dindo classification system.
Verify whether minimally invasive approaches ensure the same effectiveness than open surgery. (Overall survival.) | Assessment at 1, 3, 5 years from surgery.
  Overall survival.
Compare the three treatment arms in terms of tumor recurrence after treatment. (Disease-free survival) | Assessment at 1, 3, 5 years from surgery.
  Disease-free survival.

SECONDARY OUTCOMES:
Verify the safety of intracorporeal anastomosis in comparison with extracorporeal anastomosis. (Anastomotic leakage) | Assessment during an average period of 10 days after surgery.
  Anastomotic leakage.
Compare the intracorporeal anastomosis with the extracorporeal anastomosis to evaluate post-operative recovery. (Days of hospitalization after surgery until discharge.) | Assessment during an average period of 10 days after surgery.
  Days of hospitalization after surgery until discharge.
Verify whether robotic gastrectomy, compared with laparoscopic or open techniques, is capable of improving postoperative surgical stress. (Granulocyte-to-lymphocyte ratio.) | Assessment during an average period of 10 days after surgery.
  Granulocyte-to-lymphocyte ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Amilcare Parisi, MD, Principal Investigator — Azienda Ospedaliera S. Maria di Terni
Locations (1):
- Department of Digestive Surgery, St. Mary's Hospital, University of Perugia, Terni, Italy

REFERENCES:
- [Background] Vinuela EF, Gonen M, Brennan MF, Coit DG, Strong VE. Laparoscopic versus open distal gastrectomy for gastric cancer: a meta-analysis of randomized controlled trials and high-quality nonrandomized studies. Ann Surg. 2012 Mar;255(3):446-56. doi: 10.1097/SLA.0b013e31824682f4. PMID 22330034
- [Background] Alimoglu O, Atak I, Eren T. Robot-assisted laparoscopic (RAL) surgery for gastric cancer. Int J Med Robot. 2014 Sep;10(3):257-62. doi: 10.1002/rcs.1566. Epub 2013 Dec 23. PMID 24375986
- [Background] Shen WS, Xi HQ, Chen L, Wei B. A meta-analysis of robotic versus laparoscopic gastrectomy for gastric cancer. Surg Endosc. 2014 Oct;28(10):2795-802. doi: 10.1007/s00464-014-3547-1. Epub 2014 May 2. PMID 24789136
- [Background] Marano A, Choi YY, Hyung WJ, Kim YM, Kim J, Noh SH. Robotic versus Laparoscopic versus Open Gastrectomy: A Meta-Analysis. J Gastric Cancer. 2013 Sep;13(3):136-48. doi: 10.5230/jgc.2013.13.3.136. Epub 2013 Sep 30. PMID 24156033
- [Background] Liao G, Chen J, Ren C, Li R, Du S, Xie G, Deng H, Yang K, Yuan Y. Robotic versus open gastrectomy for gastric cancer: a meta-analysis. PLoS One. 2013 Dec 3;8(12):e81946. doi: 10.1371/journal.pone.0081946. eCollection 2013. PMID 24312610
- [Background] Hyun MH, Lee CH, Kim HJ, Tong Y, Park SS. Systematic review and meta-analysis of robotic surgery compared with conventional laparoscopic and open resections for gastric carcinoma. Br J Surg. 2013 Nov;100(12):1566-78. doi: 10.1002/bjs.9242. PMID 24264778
- [Derived] Desiderio J, Jiang ZW, Nguyen NT, Zhang S, Reim D, Alimoglu O, Azagra JS, Yu PW, Coburn NG, Qi F, Jackson PG, Zang L, Brower ST, Kurokawa Y, Facy O, Tsujimoto H, Coratti A, Annecchiarico M, Bazzocchi F, Avanzolini A, Gagniere J, Pezet D, Cianchi F, Badii B, Novotny A, Eren T, Leblebici M, Goergen M, Zhang B, Zhao YL, Liu T, Al-Refaie W, Ma J, Takiguchi S, Lequeu JB, Trastulli S, Parisi A. Robotic, laparoscopic and open surgery for gastric cancer compared on surgical, clinical and oncological outcomes: a multi-institutional chart review. A study protocol of the International study group on Minimally Invasive surgery for GASTRIc Cancer-IMIGASTRIC. BMJ Open. 2015 Oct 19;5(10):e008198. doi: 10.1136/bmjopen-2015-008198. PMID 26482769